CLINICAL TRIAL: NCT03488680
Title: Effectiveness of Behavior Change Communication on Optimal Complementary Feeding Through Community Level Actors in Improving Feeding Practices, Nutritional and Health Status of Infants in West Gojjam Zone, Northwest Ethiopia
Brief Title: Effectiveness of Behavior Change Communication in Improving Feeding Practices, Nutritional and Health Status of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Chalachew Abiyu, Principal investigator, Jimma University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RP144107
Record Dates: First submitted 2016-06-14; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Feeding Behavior; Nutritional Status; Morbidity
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Behavior change communication
  Interventions: Behavioral: Behavior change communication
- Control group (No Intervention): No Behavior change communication

INTERVENTIONS:
Behavioral: Behavior change communication — Behavior change communication about optimal complementary feeding
  Arms: Intervention group

SUMMARY:
Child under nutrition is a major risk factor for ill health and mortality, contributes substantially to the burden of disease in low-income and middle-income countries and is associated with close to half of all child deaths. The prevalence of both underweight and stunting is highest in Africa and South-Central Asia. Ethiopia is one of the poorest countries in Sub- Saharan Africa, and child malnutrition is a serious public health problem where the rates for stunting (40%), underweight (25%) and wasting (9%) among children under 5 years are among the highest in the world.

Globally, about 40% of child mortality less than two years is associated with inappropriate feeding practices. Optimal breastfeeding and appropriate complementary feeding could prevent 13% and 6% under-five mortality, respectively. Over two third of malnutrition is associated with inappropriate feeding practices during the first year of life.

The first two years of life provides a critical window of opportunity for ensuring appropriate growth and development of children from generation to generation through optimal feeding. Hence, the objective of this study to evaluate the effectiveness of behavior change communication on optimal complementary feeding through community level actors in improving feeding practice, health and nutritional status of infants.

A cluster-randomized controlled trial which was conducted in West Gojjam Zone, Northwest Ethiopia from May 9, 2016 to October, 2017. Behavior change communication on complementary feeding was conducted in the intervention kebeles/villages for 8 months. A validated interviewer administered structured questionnaire was used for collecting information on the study subjects both at the baseline and after intervention. Data will be checked, coded and double entered using EPI info and exported to SPSS version 21 for statistical analysis.

The output of the study findings could be useful for health and nutrition policy makers and other concerned bodies in decision making and to design effective intervention strategies to improve feeding practices thus mitigating child malnutrition and improving their health and growth. The total budget needed to conduct the study is 7,000 US dollar.

DETAILED DESCRIPTION:
Globally, about 40% of death children less than two years is associated with inappropriate feeding practices. Optimal breastfeeding and appropriate complementary feeding could prevent 13% and 6% under-five mortality, respectively. Over two third of malnutrition is associated with inappropriate feeding practices during the first year of life.

Every day, 3000-4000 infants die in the developing world from diarrhea and acute respiratory infections because they are given inadequate amounts of breast milk. More than 10 million children die each year in sub- Saharan Africa and South Asia. A major contributor to their deaths is poor breastfeeding practice. The risk of death from diarrhea of partially breastfed infants 0 - 6 months of age was 8.6 times the risk for exclusively breastfed children.

Infant and young feeding practices for infant and young children worldwide are not optimal. It is only 34.8% of infants are exclusively breastfed worldwide. Complementary foods are often introduced too early or too late and are often nutritionally inadequate or unsafe. Only about 39% of infants in the developing countries, 25% in Africa are exclusively breastfed for the first six months and 6% of infants in developing countries are never breastfed.

A wide range of harmful infant and young child feeding practices were documented in Ethiopia. According to EDHS of 2011, 52% of infants started breastfeeding within one hour of birth and exclusive breastfeeding during the first six months with the 4.2 months mean duration of exclusive breastfeeding. About half (49%) of children aged 6-8 months consumed solid, semi-solid, or soft foods and 5% of children were fed minimum dietary diversity and 4% of children fed minimum meal frequency per day while 96% of children continued breastfeeding at one year, and 82% continued at 2 year. Only 4% of children 6 - 23 months living with their mothers are fed in accordance with infant and young child feeding practices and 66% children under the age of two receive age-appropriate breastfeeding. Overall, nearly three children in every ten (27%) are given prelacteal feeds within the first three days of life.

In Amhara region, 38% of infants started breastfeeding within one hour of birth while only 2% and 34% of children 6-24 months were fed according to the minimum standards with respect to food diversity (four or more food groups) and meal frequency.

Sub-optimal infant and young child feeding practices are associated with caretakers' poor knowledge, lack of information and being restricted by traditional beliefs. It is essential to give caregivers necessary knowledge and information to alter their inappropriate feeding behaviors. Promotion of appropriate feeding practices, therefore, is fundamentally important in reducing child malnutrition and mortality and, thus, for achieving MDG 1. In order to sustain the gains made by promoting exclusive breastfeeding for the first six months of life, interventions need to extend into the second half of infancy and beyond. This could be ensured by enabling caregivers to appropriately feed their children with safe and adequate complementary foods while maintaining frequent breastfeeding.

Several efforts to improve the feeding status of the infant and young children have been carried out at different times. The Ethiopian government developed the infant and young child feeding guideline in 2004 following WHO recommendations of global strategy for feeding infants and young children for proper nutrition & health. Community based nutrition program was also designed to build upon the HEP packages and implemented in all agrarian regions of Ethiopia. However, these efforts have failed to bring about substantive and sustainable changes leading to improvement of infant and young child feeding practices since efforts (nutrition actions) were not based on the evidence on existing feeding practices and what works and what does not. Moreover, the health extension workers were not effectively networked with the community volunteers, work load for health extension workers and lack of training and supervision outcomes could factor their effects on the feeding practices.

As a result, the problem of stunting has remained pervasively high in the country. The government has designed an accelerated stunting reduction program under the revised national nutrition program. Moreover the Federal Ministry of Health has made reduction of child malnutrition in Ethiopia a priority flagship program under the commitment to the Seqota declaration, which states zero level hunger among under two children by 2030. Therefore, the aim of this study is to evaluate the effectiveness of behavior change communication on optimal complementary feeding through community level actors in improving feeding practice, nutrition and health status of infants.

ELIGIBILITY:
Inclusion Criteria:

* All infants aged 0-6 months at the time of baseline survey,
* Residents in the sampled villages

Exclusion Criteria:

* Mother who are ill and unable to communicate
* Infants with birth defects, impaired feeding and ill at the time of baseline survey.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 630 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Linear growth | 8 months of intevention
  Increase in linear growth (cm) after intervention

SECONDARY OUTCOMES:
Dietary diversity score | 8 months of intervention
  Dietary diversity score ranges from 1-7; dietary diversity score of greater than or equal to 4 will be considered as optimal.
Health status | 8 months of intervention
  Any form of morbidity in the last two weeks before the study
Time of initiation of complementary food | 8 months of intervention
  Time of initiation of complementary food after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chalachew Abiyu, MSc, Principal Investigator — Jimma University, Jimma, Ethiopia
Locations (1):
- Jimma University, Jimma, Ethiopia

REFERENCES:
- [Background] Sun J, Dai Y, Zhang S, Huang J, Yang Z, Huo J, Chen C. Implementation of a programme to market a complementary food supplement (Ying Yang Bao) and impacts on anaemia and feeding practices in Shanxi, China. Matern Child Nutr. 2011 Oct;7 Suppl 3(Suppl 3):96-111. doi: 10.1111/j.1740-8709.2011.00353.x. PMID 21929638
- [Derived] Ayalew CA, Belachew T. Effect of complementary feeding behaviour change communication delivered through community-level actors on infant growth and morbidity in rural communities of West Gojjam Zone, Northwest Ethiopia: A cluster-randomized controlled trial. Matern Child Nutr. 2021 Jul;17(3):e13136. doi: 10.1111/mcn.13136. Epub 2021 Jan 6. PMID 33403819
- [Derived] Abiyu C, Belachew T. Effect of complementary feeding behavior change communication delivered through community-level actors on the time of initiation of complementary foods in rural communities of West Gojjam zone, Northwest Ethiopia: a cluster-randomized controlled trial. BMC Pediatr. 2020 Nov 5;20(1):509. doi: 10.1186/s12887-020-02396-z. PMID 33153434
- [Derived] Abiyu C, Belachew T. Effect of complementary feeding behavior change communication delivered through community-level actors on dietary adequacy of infants in rural communities of West Gojjam Zone, Northwest Ethiopia: A cluster-randomized controlled trial. PLoS One. 2020 Sep 3;15(9):e0238355. doi: 10.1371/journal.pone.0238355. eCollection 2020. PMID 32881945
- See also: Olinelibray in pdf version — http://onlinelibrary.wiley.com/doi/10.1111/j.1740-8709.2011.00353.x/epdf